CLINICAL TRIAL: NCT02604017
Title: A Randomized, Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Adults With Chronic Hepatitis C Virus Genotype 1 Infection (ENDURANCE-1)
Brief Title: A Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Subjects With Genotype 1 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-590; 2015-002087-17 (EudraCT Number)
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C; Hepatitis C Virus; HCV
Keywords: HCV GT1; Non-cirrhotic; RBV Free; Without cirrhosis; Chronic Hepatitis C; Hepatitis C Genotype 1 (GT1); IFN free; Hepatitis C; Ribavirin Free; Interferon (IFN) Free; HCV; Hepatitis C virus; DAA
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABT-493/ABT-530 for 12 weeks (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 12 weeks.
  Interventions: Drug: ABT-493/ABT-530
- ABT-493/ABT-530 for 8 weeks (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 8 weeks.
  Interventions: Drug: ABT-493/ABT-530

INTERVENTIONS:
Drug: ABT-493/ABT-530 — Tablet; ABT-493 coformulated with ABT-530
  Other Names: ABT-493 also known as glecaprevir; ABT-530 also known as pibrentasvir; MAVYRET

SUMMARY:
This study seeks to evaluate the efficacy and safety of ABT-493/ABT-530 in participants with Genotype 1 hepatitis C virus infection without cirrhosis

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age at time of screening.
* Screening laboratory result indicating hepatitis C virus (HCV) genotype 1 (GT1) infection.
* Chronic HCV infection.
* Subject must be HCV treatment-naïve (i.e., patient has never received a single dose of any approved or investigational regimen) or treatment-experienced (has failed prior interferon [IFN] or pegylated IFN (pegIFN) with or without ribivarin (RBV), or sofosbuvir (SOF) plus RBV with or without pegIFN therapy).
* Subjects must be non-cirrhotic.

Additional Inclusion Criteria for HCV GT1/human immununovirus type 1 (HIV-1) co-infected patients:

* HIV-1 antiretroviral treatment (ART) naïve with CD4 ≥ 500 cells/mm3 (or CD4+ % ≥ 29%) at Screening and plasma HIV-1 RNA <1,000 copies/mL at Screening and at least once during the 12 months prior to Screening.

OR

* On a stable, qualifying HIV-1 ART regimen for at least 8 weeks prior to screening, with CD4 ≥ 200 cells/mm3 (or CD4+ % ≥14%) at Screening and plasma HIV-1 RNA < LLOQ at Screening and at least once during the 12 months prior to Screening.

Exclusion Criteria:

* History of severe, life-threatening or other significant sensitivity to any excipients of the study drugs.
* Female who is pregnant, planning to become pregnant during the study or breastfeeding; or male whose partner is pregnant or planning to become pregnant during the study.
* Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
* Positive test result at Screening for hepatitis B surface antigen (HBsAg).
* HCV genotype performed during screening indicating co-infection with more than one HCV genotype.
* Chronic HIV type 2 (HIV-2) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

REFERENCES:
- [Background] Zeuzem S, Foster GR, Wang S, Asatryan A, Gane E, Feld JJ, Asselah T, Bourliere M, Ruane PJ, Wedemeyer H, Pol S, Flisiak R, Poordad F, Chuang WL, Stedman CA, Flamm S, Kwo P, Dore GJ, Sepulveda-Arzola G, Roberts SK, Soto-Malave R, Kaita K, Puoti M, Vierling J, Tam E, Vargas HE, Bruck R, Fuster F, Paik SW, Felizarta F, Kort J, Fu B, Liu R, Ng TI, Pilot-Matias T, Lin CW, Trinh R, Mensa FJ. Glecaprevir-Pibrentasvir for 8 or 12 Weeks in HCV Genotype 1 or 3 Infection. N Engl J Med. 2018 Jan 25;378(4):354-369. doi: 10.1056/NEJMoa1702417. PMID 29365309
- [Derived] Brown A, Welzel TM, Conway B, Negro F, Brau N, Grebely J, Puoti M, Aghemo A, Kleine H, Pugatch D, Mensa FJ, Chen YJ, Lei Y, Lawitz E, Asselah T. Adherence to pan-genotypic glecaprevir/pibrentasvir and efficacy in HCV-infected patients: A pooled analysis of clinical trials. Liver Int. 2020 Apr;40(4):778-786. doi: 10.1111/liv.14266. Epub 2019 Oct 18. PMID 31568620
- [Derived] Back D, Belperio P, Bondin M, Negro F, Talal AH, Park C, Zhang Z, Pinsky B, Crown E, Mensa FJ, Marra F. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic HCV infection and psychiatric disorders: An integrated analysis. J Viral Hepat. 2019 Aug;26(8):951-960. doi: 10.1111/jvh.13110. Epub 2019 May 20. PMID 30977945
- [Derived] Gane E, Poordad F, Zadeikis N, Valdes J, Lin CW, Liu W, Asatryan A, Wang S, Stedman C, Greenbloom S, Nguyen T, Elkhashab M, Worns MA, Tran A, Mulkay JP, Setze C, Yu Y, Pilot-Matias T, Porcalla A, Mensa FJ. Safety and Pharmacokinetics of Glecaprevir/Pibrentasvir in Adults With Chronic Genotype 1-6 Hepatitis C Virus Infections and Compensated Liver Disease. Clin Infect Dis. 2019 Oct 30;69(10):1657-1664. doi: 10.1093/cid/ciz022. PMID 30923816
- [Derived] Naganuma A, Chayama K, Notsumata K, Gane E, Foster GR, Wyles D, Kwo P, Crown E, Bhagat A, Mensa FJ, Otani T, Larsen L, Burroughs M, Kumada H. Integrated analysis of 8-week glecaprevir/pibrentasvir in Japanese and overseas patients without cirrhosis and with hepatitis C virus genotype 1 or 2 infection. J Gastroenterol. 2019 Aug;54(8):752-761. doi: 10.1007/s00535-019-01569-7. Epub 2019 Mar 13. PMID 30868245
- [Derived] Foster GR, Dore GJ, Wang S, Grebely J, Sherman KE, Baumgarten A, Conway B, Jackson D, Asselah T, Gschwantler M, Tomasiewicz K, Aguilar H, Asatryan A, Hu Y, Mensa FJ. Glecaprevir/pibrentasvir in patients with chronic HCV and recent drug use: An integrated analysis of 7 phase III studies. Drug Alcohol Depend. 2019 Jan 1;194:487-494. doi: 10.1016/j.drugalcdep.2018.11.007. Epub 2018 Nov 24. PMID 30529905
- [Derived] Flamm S, Reddy KR, Zadeikis N, Hassanein T, Bacon BR, Maieron A, Zeuzem S, Bourliere M, Calleja JL, Kosloski MP, Oberoi RK, Lin CW, Yu Y, Lovell S, Semizarov D, Mensa FJ. Efficacy and Pharmacokinetics of Glecaprevir and Pibrentasvir With Concurrent Use of Acid-Reducing Agents in Patients With Chronic HCV Infection. Clin Gastroenterol Hepatol. 2019 Feb;17(3):527-535.e6. doi: 10.1016/j.cgh.2018.07.003. Epub 2018 Sep 10. PMID 30012435
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 35-day screening period.
Period: Overall Study
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Started (Intent-to-treat population: all participants who received at least 1 dose of study drug.) | 352 | 351
Completed | 346 | 343
Not Completed | 6 | 8
Not completed — Withdrew Consent | 0 | 2
Not completed — Lost to Follow-up | 5 | 6
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug (ITT population).
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks | Total
Number analyzed (Participants) | 352 | 351 | 703
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.27 (11.62) | 51.58 (11.90) | 50.93 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 184 | 360
  Male | 176 | 167 | 343

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) in Mono-infected Hepatitis C Virus Genotype 1 (HCV GT1), Direct-acting Antiviral Agent (DAA) Naïve Participants in the 12-Week Treatment Arm
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug. The primary efficacy endpoint was noninferiority of the percentage of participants who achieved SVR12 in the 12-week treatment group compared with the historical control rate for HCV GT1 subjects who are treatment-naïve or treated with pegylated-interferon alfa-2a or alfa-2b and ribavirin (pegIFN/RBV).
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants in the ITT population who were mono-infected HCV GT1, DAA-naïve; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-493/ABT-530 for 12 Weeks
Number analyzed (Participants) | 332
percentage of participants | 99.7
Statistical Analysis 1: Comparison: ABT-493/ABT-530 for 12 Weeks; Based on a 2-sided significance level of 0.05 and an underlying rate of ≥97% in the 12-week arm, 270 participants provides >90% power to demonstrate noninferiority of the 12-week arm to the historical control rate for HCV GT1 subjects who are treatment-naïve or treated with pegIFN/RBV (based on the normal approximation of a single binomial proportion in a one-sample test for superiority); Test type: Non-Inferiority — The noninferiority of the rate of SVR12 for the 12-week treatment group as compared with the historical rate was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the percentage of participants with SVR12 must exceed 91% to achieve noninferiority; Percentage of Participants = 99.7, 95% CI 2-sided [99.1 to 100.0]

2. Primary Outcome: Percentage of Participants With SVR12: Noninferiority of 8-Week Arm to 12-Week Arm in Mono-infected HCV GT1, DAA-Naïve Participants, Excluding Those Who Discontinued/Experienced Virologic Failure by Week 8 or Had No HCV RNA Value at Week 12 or Later
Description: SVR12 was defined as plasma HCV RNA level <LLOQ 12 weeks after the last dose of study drug. The primary efficacy endpoint was noninferiority of the percentage of mono-infected HCV GT1, DAA-naïve participants (excluding those who discontinued/experienced virologic failure by Week 8 or had no HCV RNA value at Week 12 or later) who achieved SVR12 in the 8-week treatment arm compared with the 12-week treatment arm.
Time Frame: 12 weeks after last actual dose of study drug
Population: All participants in the ITT population who were mono-infected HCV GT1 DAA-naïve (excluding those who discontinued/experienced virologic failure by Week 8 or had no HCV RNA value at Week 12 or later); participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Number analyzed (Participants) | 331 | 332
percentage of participants | 100.0 [98.9 to 100.0] | 100 [98.9 to 100.0]
Statistical Analysis 1: Comparison: ABT-493/ABT-530 for 12 Weeks vs ABT-493/ABT-530 for 8 Weeks; Based on a 2-sided significance level of 0.05 and an -5% noninferiority margin and an underlying rate of ≥97% in the 8-week arm (270 participants) and ≥97% in the 12-week arm (270 participants) provides >90% power to demonstrate noninferiority of the 8-week arm to the 12-week arm; Test type: Non-Inferiority — The noninferiority of the rate of SVR12 for the 8-week treatment group as compared with the 12-week treatment group was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the difference in percentage of participants with SVR12 (8-week group minus 12-week group) must be above -5% to achieve noninferiority; Difference in Percentage of Participants = 0.0, 95% CI 2-sided [-1.1 to 1.1]

3. Primary Outcome: Percentage of Participants With SVR12: Noninferiority of 8-Week Treatment Arm to 12-Week Treatment Arm in Mono-infected HCV GT1, DAA-Naïve Participants
Description: SVR12 was defined as plasma HCV RNA level <LLOQ 12 weeks after the last dose of study drug. The primary efficacy endpoint was noninferiority of the percentage of mono-infected HCV GT1, DAA-naïve participants who achieved SVR12 in the 8-week treatment arm compared with the 12-week treatment arm.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Number analyzed (Participants) | 332 | 335
percentage of participants | 99.7 [99.1 to 100.0] | 99.1 [98.1 to 100.0]
Statistical Analysis 1: Comparison: ABT-493/ABT-530 for 12 Weeks vs ABT-493/ABT-530 for 8 Weeks; Based on a 2-sided significance level of 0.05 and a -5% noninferiority margin, and an underlying rate of ≥97% in the 8-week arm (270 participants) and ≥97% in the 12-week arm (270 participants) provides >90% power to demonstrate noninferiority of the 8-week arm to the 12-week arm; Test type: Non-Inferiority — The noninferiority of the rate of SVR12 for the 8-week treatment group as compared with the 12-week treatment group was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the difference in percentage of participants with SVR12 must be above -5% to achieve noninferiority; Difference in Percentage of Participants = -0.6, 95% CI 2-sided [-1.8 to 0.6]

4. Secondary Outcome: Percentage of Participants With SVR12 in Mono-infected HCV GT1 Participants
Description: SVR12 was defined as plasma HCV RNA level <LLOQ 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after last actual dose of study drug
Population: All participants in the ITT population who were mono-infected HCV GT1; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Number analyzed (Participants) | 334 | 336
percentage of participants | 99.7 [98.3 to 99.9] | 99.1 [97.4 to 99.7]

5. Secondary Outcome: Percentage of Participants With SVR12
Description: SVR12 was defined as plasma HCV RNA level <LLOQ 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after last actual dose of study drug
Population: All participants in the ITT population; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Number analyzed (Participants) | 352 | 351
percentage of participants | 99.7 [98.4 to 99.9] | 99.1 [97.5 to 99.7]

6. Secondary Outcome: Percentage of Participants With SVR12 in Co-infected HCV GT1/Human Immunodeficiency Virus Type 1 (HIV-1) Participants
Description: SVR12 was defined as plasma HCV RNA level <LLOQ 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after last actual dose of study drug
Population: All participants in the ITT population who were co-infected HCV GT1/HIV-1; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Number analyzed (Participants) | 18 | 15
percentage of participants | 100.0 [82.4 to 100.0] | 100.0 [79.6 to 100.0]

7. Secondary Outcome: Percentage of Participants With SVR12 in HCV GT1-infected, Prior Sofosbuvir (SOF) Treatment-Experienced Participants
Description: SVR12 was defined as plasma HCV RNA level <LLOQ 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after last actual dose of study drug
Population: All participants in the ITT population who were HCV GT1-infected, prior SOF-treatment experienced; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Number analyzed (Participants) | 2 | 1
percentage of participants | 100.0 [34.2 to 100.0] | 100.0 [20.7 to 100.0]

8. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed increase of >1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline HCV RNA during treatment; confirmed HCV RNA ≥100 IU/mL after HCV RNA <LLOQ during treatment, or HCV RNA ≥LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: Treatment Weeks 1, 2, 4, 8 (end of treatment for 8-week treatment arm), and 12 (end of treatment for 12-week treatment arm) or premature discontinuation from treatment
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Number analyzed (Participants) | 352 | 351
percentage of particpants | 0.0 [0.0 to 1.1] | 0.3 [0.1 to 1.6]

9. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure in Mono-infected HCV GT1, DAA-Naïve Participants
Description: as for outcome 8
Time Frame: as for outcome 8
Population: All participants in the ITT population who were mono-infected HCV GT1, DAA-naïve.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Number analyzed (Participants) | 332 | 335
percentage of participants | 0.0 [0.0 to 1.1] | 0.3 [0.1 to 1.7]

10. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels <LLOQ at the end of treatment, excluding reinfection.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Number analyzed (Participants) | 352 | 349
percentage of participants | 0.0 [0.0 to 1.1] | 0.0 [0.0 to 1.1]

11. Secondary Outcome: Percentage of Participants With Post-treatment Relapse in Mono-infected HCV GT1, DAA-Naïve Participants
Description: as for outcome 10
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants in the ITT population who were mono-infected HCV GT1, DAA-naïve, received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Number analyzed (Participants) | 332 | 333
percentage of participants | 0.0 [0.0 to 1.1] | 0.0 [0.0 to 1.1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and TESAEs are defined as any AE or SAE with an onset or worsening date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ABT-493/ABT-530 for 12 Weeks | ABT-493/ABT-530 for 8 Weeks
Serious Adverse Events (participants affected / at risk) | 4/352 | 5/351
Other Adverse Events (participants affected / at risk) | 130/352 | 133/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-493/ABT-530 for 12 Weeks (N=352) | ABT-493/ABT-530 for 8 Weeks (N=351)
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 0
ARTERIAL INJURY (Injury, poisoning and procedural complications) | 0 | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-493/ABT-530 for 12 Weeks (N=352) | ABT-493/ABT-530 for 8 Weeks (N=351)
NAUSEA (Gastrointestinal disorders) | 29 | 19
FATIGUE (General disorders) | 43 | 31
NASOPHARYNGITIS (Infections and infestations) | 31 | 22
HEADACHE (Nervous system disorders) | 62 | 68
INSOMNIA (Psychiatric disorders) | 15 | 21
PRURITUS (Skin and subcutaneous tissue disorders) | 17 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.